CLINICAL TRIAL: NCT05956808
Title: Phonak Behind-The-Ear Quality Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-12872
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: This investigation model is a cross-over design, randomized, and is single-blinded.
Who Masked: Participant
Masking Description: Participants will be blinded as to which hearing device they are wearing during lab testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- New BTE hearing aid first, then legacy BTE hearing aid (Experimental): All participants who complete speech intelligibility testing and subjective listening effort ratings with both devices, first with the new hearing aid, and then with the legacy hearing aid.
  Interventions: Device: Phonak Naida BTE hearing aid; Device: Phonak Naida legacy BTE hearing aid
- Legacy BTE hearing aid first, then new BTE hearing aid (Experimental): All participants who complete speech intelligibility testing and subjective listening effort ratings with both devices, first with the new hearing aid, and then with the legacy hearing aid.
  Interventions: Device: Phonak Naida BTE hearing aid; Device: Phonak Naida legacy BTE hearing aid

INTERVENTIONS:
Device: Phonak Naida BTE hearing aid — Newest generation of ultra-power Phonak BTE hearing aids
Device: Phonak Naida legacy BTE hearing aid — Previous model/generation of the Naida BTE hearing aid

SUMMARY:
Subjective listening effort and objective speech intelligibility will be evaluated with a new generation of a Phonak BTE (Behind-The-Ear) hearing aid.

DETAILED DESCRIPTION:
Speech intelligibility performance will be measured with a new generation BTE hearing aid and compared to a legacy hearing aid in adults with severe to profound hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Severe to profound hearing loss (4 frequency Pure Tone Average 65-94 dB)
* 18+ years old
* Good written and spoken English language skills
* Able to fill in a questionnaire conscientiously
* Experienced hearing aid user
* Able to produce a reliable hearing test result
* Able to describe listening impressions/experiences and the use of the hearing aids

Exclusion Criteria:

* Not willing to test the hearing aids
* Has auricle deformities that prevents secure placement of the hearing aids
* Has limited mobility and is not able to attend the appointments
* Not willing to wear the hearing aids for at least 8 hours per day
* Known hypersensitivity or allergy with synthetic materials
* Self reports symptoms of vertigo, dizziness, fluctuating hearing loss
* Hints of psychological problems
* Suffers from acute tinnitus in either one or both ears (occurrence less than 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Speech in Noise Test | Day 14 of the study
  Sentences are presented to either the left or right side of the participant's head through a speaker that is 1 meter away. Background noise is presented through the remaining seven speakers that are arranged in a circular pattern around the participant. The sentences are presented at varying levels which may be both louder and softer than the fixed level of noise. The SNR50 is the Signal to Noise Ratio (SNR) at which the participant can repeat 50% of the words correctly. For example, an SNR50 of +3 means that the participant repeated 50% of the words back correctly when the sentences were presented at a level that was 3 dB louder than the noise. Lower SNR50 scores indicate better performance.
Subjective measure of listening effort | Day 14 of the study
  A rating scale will be given to the participants following the Speech in Noise Test in which they will rate their perceived listening effort during the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Phonak Audiology Research Center, Aurora, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared outside of Sonova research departments.